CLINICAL TRIAL: NCT02858011
Title: The Effect of a Cash Transfer Program and Preventive Nutrition Packages on Household Welfare and Child Nutritional Status in Mali
Acronym: Jigisemejiri
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Implementation management committee of the Jigisemejiri program (Ministry of Economics and Finance, Government of Mali) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-26-PHND-M
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Poverty; Child Malnutrition
Keywords: behavior change communication; cash transfer; household welfare; child nutrition status
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Child Nutritional Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control and comparison group -cash transfer program (Active Comparator): The program is implemented during 48 months. During the first 36 months the control group does not receive any intervention. During the last 12 months eligible beneficiaries receive cash transfer and accompanying information sessions on health, child nutrition, household economics every three months (identical to experimental group).
  Interventions: Other: Cash distribution during the last 12 months; Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during the last 12 months
- Jigisemejiri cash transfer program (Experimental): Unconditional cash is distributed every 3 months to beneficiaries of the Jigisemejiri program. During cash handouts, information sessions on health, child nutrition, households economics and education are organized by local NGOs.
  Interventions: Other: Cash distribution during first 36 months; Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during first 36 months
- Jigisemejiri - Preventive Nutrition packages (Experimental): Households belonging to the experimental group who previously received Cash transfer and information sessions on health, child nutrition, households economics and education for 36 months, with children and/or pregnant/lactating women receiving rations of fortified flour (PNP) during the last 12 months of the project
  Interventions: Other: Cash distribution during first 36 months; Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during first 36 months; Dietary Supplement: Preventive Nutrition Packages during last 12 months
- Control and comparison group - Preventive Nutrition packages (Active Comparator): Households belonging to the experimental group who previously received Cash transfer and information sessions on health, child nutrition, households economics and education for 36 months, with children and/or pregnant/lactating women
  Interventions: Other: Cash distribution during first 36 months; Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during first 36 months

INTERVENTIONS:
Other: Cash distribution during first 36 months — Three-monthly distribution of Cash (30,000 FCFA/trimester) to households that are beneficiary of the Jigisemejiri program.
  Arms: Control and comparison group - Preventive Nutrition packages; Jigisemejiri - Preventive Nutrition packages; Jigisemejiri cash transfer program
Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during first 36 months — Large group gatherings of cash beneficiaries are organized in parallel to the cash distributions. During these meetings, local NGOs present and discuss a topic related to health, child nutrition, household economics or education.
  Arms: Control and comparison group - Preventive Nutrition packages; Jigisemejiri - Preventive Nutrition packages; Jigisemejiri cash transfer program
Dietary Supplement: Preventive Nutrition Packages during last 12 months — Fortified flour supplements for children (Supercereal Plus)and pregnant/lactating mothers (super Cereal)
  Arms: Jigisemejiri - Preventive Nutrition packages
Other: Cash distribution during the last 12 months — Three-monthly distribution of Cash (30,000 FCFA/trimester) to households that are beneficiary of the Jigisemejiri program.
  Arms: Control and comparison group -cash transfer program
Behavioral: Accompanying information sessions on health, child nutrition, household economics and education during the last 12 months — Large group gatherings of cash beneficiaries are organized in parallel to the cash distributions. During these meetings, local NGOs present and discuss a topic related to health, child nutrition, household economics or education.
  Arms: Control and comparison group -cash transfer program

SUMMARY:
In the last two decades, cash transfer (CT) programs have emerged as a popular approach to long-term poverty alleviation. While the main goal of cash transfer programs is to reduce poverty, they also have the potential to improve many development outcomes, such as health and education.

While many studies, mainly in Latin America and Asia, have investigated the impacts of CTs on poverty and food security and have, for the most part, found positive impacts, less is known about the impacts of CTs in Africa south of the Sahara, and, in particular, West Africa. Moreover, despite the fact that cash transfers have been shown to lead to decreases in poverty, improvements in household food security, and increases in health service utilization, impacts on children's nutritional status (including anthropometric measures) are generally small (Manley, Gitter, and Slavchevska 2013). Consequently, policymakers and governments are left with the question of how to design social safety nets, such as cash transfers, to achieve greater impact on diet quality, health, and nutrition.

The overall goal of this research is to generate evidence and knowledge on an integrated program implemented by the Government of Mali that includes a combination of cash transfers and targeted nutrition interventions. The information generated will inform program implementers and policymakers about best options to improve food security and nutrition among vulnerable groups and individuals in West Africa. Specifically, the main objectives of the research are

1. To provide evidence on the contribution of integrated social transfer programs to enhancing household welfare, food security, dietary diversity, and maternal and child nutrition in West Africa.
2. To test different features and combinations of cash transfers and targeted nutrition interventions, and assess their impact on food security and maternal and child nutrition and health outcomes in Mali.
3. To generate knowledge regarding the pathways of impact of these different program packages, identify the most effective and efficient modalities in the context of Mali, and derive lessons learned for other countries in the region.

DETAILED DESCRIPTION:
The research entails two study designs: i) a repeated cross-sectional survey (baseline, midline and endline) in a sample of 1,440 children between 6 and 24 months of age, mainly to asses the program's impact on child nutrition and health outcomes; ii) a panel study following a cohort of 2,880 children over 3 years mainly focusing on the evaluation of household welfare outcomes. The study will be conducted in the 96 communes where the Jigisemejiri program is being implemented, situated in 5 regions of Mali: Sikasso, Koulikoro, Segou, Mopti and Kayes. Data will be collected at baseline (2014, T=0), midline (2016, T=~24 months) and endline (2018, T=~48 months).

The program is implemented for 48 months. The experimental group receives the cash transfer and group counselling intervention for 36 months. During the last 12 months the experimental group does not receive any intervention. The control group receives no intervention during the first 36 months, but receives the cash transfer and group counselling during the last 12 months. In a subsample of communes from the experimental group, villages were randomized to either receive Preventive Nutrition Packages (PNP) or nothing. The impact of PNP is analyzed by comparing villages that received PNP and villages that did not receive PNP during the last 12 months of the program.

ELIGIBILITY:
Inclusion Criteria:

* Being a Household that is beneficiary of the Jigisemejiri program
* Having a child between 6 and 24 months of age

Exclusion Criteria:

* Congenital malformations that hamper anthropometric measurements

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4320 (Actual)
Dates: Start 2014-09; Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Child Height-for-age Z-score | After 24 months of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Value of household consumption | After 24 months of program implementation
  The household consumption includes food and non-food related economic consumption
Household dietary diversity | After 24 months of program implementation
  The household dietary diversity is estimated by a dietary diversity score counting food groups
Child Height-for-age Z-score | After 48 months of program implementation (only in cross-sectional survey)
  To calculate HAZ scores the 2006 WHO growth reference will be used (only in cross-sectional survey)
Value of household consumption | After 48 months of program implementation
  The household consumption includes food and non-food related economic consumption
Household dietary diversity | After 48 months of program implementation
  The household dietary diversity is estimated by a dietary diversity score counting food groups
Child Weight-for-Height Z-score | After 48 months of program implementation (only in cross-sectional survey)
  To calculate WHZ scores the 2006 WHO growth reference will be used (only in cross-sectional survey)

SECONDARY OUTCOMES:
Child Weight-for-height Z-score | After 24 months of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Prevalence of child wasting | After 24 months and 48 months (only in cross-sectional survey) of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Prevalence of child stunting | After 24 months and 48 months (only in cross-sectional survey) of program implementation
  To calculate WHZ scores the 2006 WHO growth reference will be used
Child hemoglobin concentration | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Prevalence of child anemia | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Body Mass Index of primary caregiver of index child | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Early child development | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Child morbidity (acute respiratory infections, fever, vomiting, diarrhea) | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Caregiver's knowledge and practices related to Infant and Young Child Feeding (IYCF), child health and hygiene | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Household assets and savings | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Educational level of Household members | After 24 months and 48 months of program implementation
Household food security | After 24 months and 48 months of program implementation
  Measured by the Household Food Insecurity Access Scale (HFIAS)
Household composition | After 24 months and 48 months of program implementation
  This entails the household size, the number of one parent households, monogamous and polygamous households, number of infants and children.
Household agricultural production | After 24 months and 48 months of program implementation
  The composition and quantity of all crops grown by the houshold over the last year is being recalled
Cognitive function of the head of household | After 24 months of program implementation
  Measured by spatial Stroop test and digit span test (forward and backward)
Well-being of household members | After 24 months and 48 months of program implementation
  Well-being is assessed by measuring stress, anxiety, psychological well-being, partner violence, marital quality, depression, occurrence of disputes and resource allocation.
Women's empowerment | After 24 months and 48 months of program implementation
  Measured by pro-WEAI instrument adapted to local context
Child dietary diversity | After 24 months and 48 months (only in cross-sectional survey) of program implementation
  Child dietary diversity is estimated by a dietary diversity score counting food groups consumed
Professional occupation of household members | After 24 months and 48 months of program implementation
  We assess if household members have different formal and informal professional occupations or main revenue generating activities between intervention and control group
Child Mid-upper Arm Circumference | After 24 months and 48 months (only in cross-sectional survey) of program implementation
Maternal hemoglobin concentration | After 48 months (only in cross-sectional survey) of program implementation
Maternal anemia | After 48 months (only in cross-sectional survey) of program implementation

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gilligan, PhD, Study Chair — IFPRI; Marie Ruel, PhD, Study Chair — IFPRI; Melissa Hidrobo, PhD, Principal Investigator — IFPRI; Shalini Roy, PhD, Principal Investigator — IFPRI; Lieven Huybregts, PhD, Principal Investigator — IFPRI
Locations (1):
- Bamako, Mali

IPD SHARING:
Plan to Share IPD: No